CLINICAL TRIAL: NCT01523652
Title: Studio Pilota Farmacocinetico-clinico Sulla Somministrazione di Eparina a Basso Peso Molecolare e Dosaggio Sierico di HGF Nelle Pazienti Operate Affette da Patologie Ginecologiche
Brief Title: Pharmacokinetic Study on the Administration of Nadroparin Dosing Serum HGF in Gynecological Patients
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliera San Giovanni Battista (Other)
Collaborators: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Paolo Zola, Prof Paolo Zola, Azienda Ospedaliera San Giovanni Battista
Other Study IDs: FRFUnito60_07
Record Dates: First submitted 2011-07-05; First posted 2012-02-01 (Estimated); Last update posted 2012-02-01 (Estimated); Status verified 2012-01

CONDITIONS: Genital Diseases, Female; Ovarian Neoplasms; Urogenital Neoplasms
MeSH Terms: conditions — Genital Diseases, Female; Ovarian Neoplasms; Urogenital Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Nadroparin/control (phase 1): patients affected by benign pelvic gynaecologic diseases were enrolled and treated with nadroparin for prophylactic anticoagulation; patients untreated with nadroparin were as control group.
- Nadroparin (phase 2): patients were enrolled among women planning gynaecological pelvic surgery and treated for 4 weeks with nadroparin for prophylactic anticoagulation. All these patients underwent laparotomy;

SUMMARY:
The purpose of this study is to determine whether HGF serum concentration might be raised in vivo by administering nadroparin given with prophylactic purpose to gynecological patients.

DETAILED DESCRIPTION:
The study consisted of two phases. In the first phase, the main HGF pharmacokinetic parameters were evaluated, comparing a group of six women treated with a single dose of calcic nadroparin to a control group of six untreated women. Venous blood was drawn in both groups at 0, 30, 60, 90, 120, 150, 180, 240, 300, 360, 480 and 720 min. In the second phase, the HGF basal and maximum concentrations were measured in 17 women, undergoing one month of calcic nadroparin daily treatment. Venous blood was drawn twice on day 1 (at 0 and 90 min after nadroparin administration), then once on days 8 and 28 (at 90 min after LMWH injection). Calcic nadroparin was given subcutaneously at 2850 IU/0.3 ml anti-Xa.

Patients' characteristics:

In the first phase, 12 patients were enrolled, 6 treated with nadroparin for prophylactic anticoagulation and another 6 untreated as the control group. The six nadroparin-group patients were affected by benign pelvic gynaecologic diseases: three requiring laparoscopy and three laparotomy.

In the control group, four were healthy women volunteers and two patients submitted to gynaecological pelvic surgery, but these women were not treated with prophylactic LMWH.

In the second phase, 17 patients were enrolled among women planning gynaecological pelvic surgery and treated for 4 weeks with nadroparin for prophylactic anticoagulation. All these patients underwent laparotomy; ten were affected by malignancy (ECOC) and seven by benign (uterine fibroma, ovarian cystadenoma) pelvic gynaecologic diseases.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years
* ECOG PS ≤ 1
* Neutrophils ≥ 1500 l -1, platelets ≥ 150,000 l -1, creatinine 0.6 to 1.2 mg dl -1, total bilirubin ≤ 1 mg dL -1, AST ≤ 35 U l-1, ALT ≤ 45 U l-1

For patients in the study group: high-moderate risk of deep vein thrombosis (for the administration of LMWH for 30 days after surgery) under general anesthesia> 30 minutes, laparoscopy + at least one risk factor (age> 40 years, obesity, varicose veins, previous episode of deep vein thrombosis and / or pulmonary thromboembolism, thrombophilia, malignancy, prolonged immobility, congestive heart failure)

Exclusion Criteria:

* severe liver and renal disease
* diabetes
* hyperlipidemia
* marked osteoporosis
* HIV infection
* ongoing treatment with: immunosuppressive therapies, contraceptives, lipid-lowering drugs, NSAIDs, antiplatelet drugs, recent acute inflammatory or infectious (<3 weeks)
* a history of allergies,
* drug possible confounding, caffeine, tobacco, ethanol (must not have been hired in the last 24 hours prior to sampling)
* high risk of bleeding: peptic ulcer, history of hemorrhagic stroke, or bleeding disorders, severe hypertension, cerebral aneurysms, arteriovenous malformations, brain metastases

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: primary care clinic gynecological patients (benign diseases, oncological diseases)
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2007-11; Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
AUC | 1 hour after nadroparin administration
  HGF serum concentration

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Zola, MD, Principal Investigator — University of Turin, Italy
Locations (1):
- ASO Ordine Mauriziano, Turin, Italy

REFERENCES:
- [Derived] Surbone A, Fuso L, Passera R, Ferrero A, Marchese C, Martino C, Luchin A, Di Renzo MF, Zola P. Daily administration of low molecular weight heparin increases Hepatocyte Growth Factor serum levels in gynaecological patients: pharmacokinetic parameters and clinical implications. BMC Res Notes. 2012 Sep 23;5:517. doi: 10.1186/1756-0500-5-517. PMID 22999213